CLINICAL TRIAL: NCT00616122
Title: Phase I/II Study of SU11248 (Sutent) in Combination With Metronomic Dosing of Cyclophosphamide and Methotrexate in Patients With Metastatic Breast Cancer
Brief Title: Sunitinib, Cyclophosphamide, and Methotrexate in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Risk to benefit ratio not acceptable
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 057519; NCI-2011-01275 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Cyclophosphamide; Methotrexate; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sunitinib, Cyclophosphamide, and Methotrexate (Experimental)
  Interventions: Drug: cyclophosphamide; Drug: methotrexate; Drug: sunitinib malate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cyclophosphamide
Drug: methotrexate
Drug: sunitinib malate
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and methotrexate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sunitinib together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of sunitinib when given together with cyclophosphamide and methotrexate to see how well they work in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of the combination of metronomic dose cyclophosphamide and methotrexate with continuous dosing sunitinib malate. (Phase I)
* To determine the time to disease progression in patients with metastatic breast cancer treated with metronomic dose chemotherapy with cyclophosphamide and methotrexate combined with continuous dosing of sunitinib malate. (Phase II)

Secondary

* To determine the response rate in patients receiving this treatment.
* To determine the duration of response in patients receiving this treatment.
* To determine the toxicity of this regimen in these patients.
* To determine the feasibility by assessment of toxicities of this regimen and number of voluntary withdrawals from the study.
* To correlate outcome measures with possible surrogate markers including serial measurements of circulating tumor cells and circulating endothelial cells.

OUTLINE: This is a dose-escalation study of sunitinib malate.

* Phase I: Patients receive oral sunitinib malate once daily. Beginning 14 days later, patients also receive oral cyclophosphamide once daily on days 1-21 and oral methotrexate twice daily on days 1, 2, 8, 9, 15, and 16. Treatment with sunitinib malate, cyclophosphamide, and methotrexate repeats every 21 days* in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients receive sunitinib malate at the maximum tolerated dose determined in phase I and cyclophosphamide and methotrexate as in phase I.

NOTE: *Course 1 includes 2 weeks of sunitinib malate alone followed by sunitinib malate, cyclophosphamide, and methotrexate for 21 days

Blood samples are collected periodically for measurement of circulating tumor cells, circulating endothelial cells, and vascular endothelial growth factor (VEGF) levels.

After completion of study treatment, patients are followed for 30 days and then every 2 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed diagnosis of breast cancer with documented progressive disease

  * Metastatic disease
* Measurable disease as defined by RECIST criteria or evaluable disease
* Must have received at least one prior chemotherapy regimen for metastatic breast cancer

  * Patients refusing all other chemotherapy for breast cancer may enroll without prior treatment
* Patients with HER2-overexpression disease must have been previously treated with trastuzumab (Herceptin®)
* Patients with stable brain metastases are eligible
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute Neutrophil Count (ANC) ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN (≤ 5 times ULN in the presence of liver metastases)
* Total bilirubin ≤ 1.5 times ULN
* Able to take oral medications and maintain hydration
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after treatment
* No severe concurrent illness including, but not limited to, any of the following:

  * Congestive heart failure
  * Significant cardiac disease
  * Uncontrolled hypertension
* Must be able to read and speak English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior treatment, including chemotherapy, hormonal therapy, trastuzumab (Herceptin®), or other targeted therapies
* Prior bevacizumab allowed if discontinued for any reason other than toxicity
* No potent inducers or inhibitors of CYP3A4 enzymes that effect the metabolism of sunitinib malate
* No prior sunitinib malate
* No other concurrent investigational therapy
* No concurrent radiotherapy
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2012-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I patients received escalating doses of sunitinib in a 3x3 design. None of the patients in the phase I study was included in phase II. Phase I patients receiving treatment at the phase II dose were included in the overall efficacy analysis of the phase II study but were not counted toward the enrollment accrual of the phase II study.
Groups:
- Phase I, Dose 1: One cycle = 21 days
  Sunitinib only (12.5 mg) for 2 weeks, followed by the addition of metronomic cyclophosphamide (50mg/day) and methotrexate (2.5mg twice a day (BID) 2 days/week).
  Patients in each cohort will be followed for at least 8 weeks (2 week lead in with sunitinib and 6 weeks of treatment with sunitinib and metronomic cyclophosphamide and methotrexate) before opening accrual to the next dose level.
- Phase I, Dose 2: One cycle = 21 days
  Sunitinib only (25 mg) for 2 weeks, followed by the addition of metronomic cyclophosphamide (50mg/day) and methotrexate (2.5mg BID 2 days/week).
  Patients in each cohort will be followed for at least 8 weeks (2 week lead in with sunitinib and 6 weeks of treatment with sunitinib and metronomic cyclophosphamide and methotrexate) before opening accrual to the next dose level.
- Phase I, Dose 3: One cycle = 21 days
  Sunitinib only (37.5 mg) for 2 weeks, followed by the addition of metronomic cyclophosphamide (50mg/day) and methotrexate (2.5mg BID 2 days/week).
  Patients in each cohort will be followed for at least 8 weeks (2 week lead in with sunitinib and 6 weeks of treatment with sunitinib and metronomic cyclophosphamide and methotrexate) before opening accrual to the next dose level.
- Phase II: * 37.5mg sunitinib during the 2-week lead-in period followed by either:
  * 37.5mg sunitinib
  * metronomic cyclophosphamide (50mg/day) and methotrexate (2.5mg BID 2 days/week)(CM)
  * 25mg sunitinib
  * metronomic CM (50mg/day)
  * methotrexate (2.5mg BID 2 days/week)
Period: Overall Study
Arm/Group | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II
Started | 4 | 7 | 10 | 11
Completed | 4 | 7 | 10 | 0
Not Completed | 0 | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib, Cyclophosphamide, and Methotrexate: Phase I patients received escalating doses of sunitinib in a 3x3 design (12.5, 25, 37.5 mg). Phase I and II patients received sunitinib for 2 weeks, followed by the addition of metronomic cyclophosphamide (50mg/day) and methotrexate (2.5mg BID 2 days/week). Phase II patients received 37.5mg sunitinib during the 2-week lead-in period followed by either 37.5mg sunitinib and metronomic CM or 25mg sunitinib and metronomic CM (dose reduction due to a protocol amendment).
Arm/Group | Sunitinib, Cyclophosphamide, and Methotrexate
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Sunitinib (Phase I)
Description: Patients in each cohort were followed for DLT for at least 8 weeks (2 week lead-in with sunitinib and 6 weeks of treatment with sunitinib and metronomic cyclophosphamide and methotrexate) before opening accrual to the next dose level. Dose limiting toxicity (DLT) defined as: 1) ≥ grade 3 anemia that does not resolve with appropriate growth factors afebrile grade 4 neutropenia that does not resolve with growth factor support after ≥ 7 days 2) grade 4 neutropenia associated with fever (1 reading of oral temperature > 38.5 degrees Celsius or 3 readings of oral temperature > 38.0 degrees Celsius in a 24 hour period) 3) ≥ grade 3 thrombocytopenia 4) ≥ grade 3 non-hematologic toxicities, except those that can be controlled to grade 2 or less with appropriate treatment.
  5) Inability to resume treatment with any of the study medications within 14 days of stopping due to treatment related toxicity.
Time Frame: 8 weeks
Measure: Number; unit: mg
Arm/Group | Sunitinib, Cyclophosphamide, and Methotrexate
Number analyzed (Participants) | 21
mg | 37.5

2. Primary Outcome: Patients With Progression-free Survival (PFS) Greater Than or Equal to 12 Weeks (Phase II)
Description: Progression defined as: 25% increase or an increase of 10 sq. cm (whichever is smaller) in the sum of products of measurable lesions over smallest sum observed (over baseline if no decrease), or appearance of any lesion which had disappeared, or clear worsening of any evaluable disease, or appearance of any new lesion/site, or failure to return for evaluation due to deteriorating condition (unless deterioration is clearly unrelated to this cancer).
Time Frame: up to 12 weeks after treatment start date
Population: Patients who received either 25mg or 37.5mg of sunitinib and were not removed from study due to voluntary withdrawal or PD prior to receiving combination sunitinib and metronomic CM chemotherapy.
Measure: Number; unit: participants
Arm/Group | Sunitinib, Cyclophosphamide, and Methotrexate
Number analyzed (Participants) | 23
participants | 7

3. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria in Solid Tumors (RECIST): Complete Response (CR): Complete disappearance of all measurable and evaluable disease. No new lesions.
  Partial Response (PR): greater than or equal to 50% decrease under baseline in the sum of the products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
  Stable: Does not qualify for complete response, partial response or progression.
Time Frame: until disease progression, up to 13 months post treatment
Measure: Number; unit: participants
Arm/Group | Sunitinib, Cyclophosphamide, and Methotrexate
Number analyzed (Participants) | 23
participants | 1

4. Secondary Outcome: Duration of Response
Description: Duration of response refers to duration of single partial response observed per Response Evaluation Criteria in Solid Tumors (RECIST):
  Complete Response (CR): Complete disappearance of all measurable and evaluable disease. No new lesions.
  Partial Response (PR): greater than or equal to 50% decrease under baseline in the sum of the products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
  Stable: Does not qualify for complete response, partial response or progression.
  Progression: 25% increase or an increase of 10 sq. cm (whichever is smaller) in the sum of products of measurable lesions over smallest sum observed (over baseline if no decrease), OR appearance of any lesion which had disappeared, or clear worsening of any evaluable disease, or appearance of any new lesion/site, or failure to return for evaluation due to deteriorating condition (unless deterioration is clearly unrelated to this cancer).
Time Frame: until disease progression up to 13 months post treatment
Population: A partial response was only reported for one patient, while a complete response was not recorded for any patients.
Measure: Number; unit: weeks
Arm/Group | Sunitinib, Cyclophosphamide, and Methotrexate
Number analyzed (Participants) | 1
weeks | 10.6

ADVERSE EVENTS:
Groups:
- Phase I, Dose 1: One cycle = 21 days
  Sunitinib only (12.5 mg) for 2 weeks, followed by the addition of metronomic cyclophosphamide (50mg/day) and methotrexate (2.5mg BID 2 days/week).
  Patients in each cohort will be followed for at least 8 weeks (2 week lead in with sunitinib and 6 weeks of treatment with sunitinib and metronomic cyclophosphamide and methotrexate) before opening accrual to the next dose level.
- Phase II: * 37.5mg sunitinib during the 2-week lead-in period followed by either:
  * 37.5mg sunitinib
  * metronomic CM (50mg/day)
  * methotrexate (2.5mg BID 2 days/week)
  or
  * 25mg sunitinib
  * metronomic CM (50mg/day)
  * methotrexate (2.5mg BID 2 days/week)
  (dose reduction due to a protocol amendment)
Arm/Group | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 1/10 | 0/11
Other Adverse Events (participants affected / at risk) | 2/4 | 6/7 | 8/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Dose 1 (N=4) | Phase I, Dose 2 (N=7) | Phase I, Dose 3 (N=10) | Phase II (N=11)
fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Dose 1 (N=4) | Phase I, Dose 2 (N=7) | Phase I, Dose 3 (N=10) | Phase II (N=11)
abdominal distention (Gastrointestinal disorders) | 0 | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0
alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 4
alkaline phosphatase increased (Investigations) | 2 | 0 | 2 | 4
allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0
alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
anal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
anemia (Blood and lymphatic system disorders) | 0 | 2 | 5 | 7
anorexia (Metabolism and nutrition disorders) | 1 | 4 | 3 | 1
anxiety (Psychiatric disorders) | 0 | 2 | 0 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
aspartate aminotransferase increased (Investigations) | 2 | 0 | 4 | 6
back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 0
blood blirubin increased (Investigations) | 0 | 0 | 2 | 2
blood urea nitrogen increased (Investigations) | 0 | 0 | 0 | 1
breast infection (Infections and infestations) | 1 | 0 | 0 | 0
bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
chills (General disorders) | 0 | 1 | 1 | 2
cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0
cold sore (Gastrointestinal disorders) | 0 | 1 | 0 | 0
constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 3
creatinine increased (Investigations) | 0 | 0 | 0 | 3
depression (Psychiatric disorders) | 0 | 0 | 1 | 1
desquamation, blistering (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
diarrhea (Gastrointestinal disorders) | 0 | 2 | 7 | 5
dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
dry eyes (Eye disorders) | 0 | 0 | 1 | 0
dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
dry mucous membrane (Gastrointestinal disorders) | 0 | 0 | 0 | 1
dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
dullness in lungs (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
dysgeusia (Gastrointestinal disorders) | 0 | 1 | 2 | 3
dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
edema limbs (General disorders) | 0 | 1 | 0 | 2
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
esophagoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
fatigue (General disorders) | 0 | 5 | 7 | 7
fever (General disorders) | 0 | 1 | 0 | 4
floaters (Eye disorders) | 0 | 0 | 1 | 0
gastroesophageal reflux disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1
gastrotitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
hand stiffness (Nervous system disorders) | 0 | 1 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 3 | 3
heavy eyelid (Eye disorders) | 0 | 1 | 0 | 0
hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
hot flashes (Vascular disorders) | 1 | 0 | 0 | 0
hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
hypertension (Vascular disorders) | 0 | 0 | 2 | 3
hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
hypochloremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
impaired LV (Cardiac disorders) | 0 | 0 | 0 | 1
insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2
jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
lightheadedness (Nervous system disorders) | 1 | 0 | 0 | 1
loss of function in right hand (Nervous system disorders) | 0 | 1 | 0 | 0
lymphocyte count decreased (Investigations) | 0 | 0 | 5 | 3
mucositis oral (Gastrointestinal disorders) | 0 | 5 | 1 | 2
myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 3
myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 2 | 5 | 4
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
neutrophil count decreased (Investigations) | 0 | 6 | 8 | 9
night sweats (Vascular disorders) | 0 | 0 | 0 | 1
non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2
numbness to chin (Nervous system disorders) | 0 | 1 | 0 | 0
oral pain (Gastrointestinal disorders) | 0 | 0 | 3 | 1
pain (General disorders) | 0 | 0 | 3 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 5
palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 4 | 3
petechia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
platelet count decreased (Investigations) | 0 | 3 | 4 | 9
pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
puffy eyelid (Eye disorders) | 0 | 1 | 0 | 0
pulsing in ear (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
rib pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
skin peeling (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
spider bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0
upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0
urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 4
warmth to chest wall (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
weight loss (Investigations) | 0 | 0 | 1 | 0
white blood cell decreased (Investigations) | 0 | 0 | 6 | 6

LIMITATIONS AND CAVEATS:
Based on published literature indicating significant toxicity and low response rate for combination sunitinib in the treatment of advanced breast cancer, the PI and Breast Oncology Site Committee closed enrollment after accrual of 32 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No